CLINICAL TRIAL: NCT02204735
Title: Timing of Meals for Weight Loss
Acronym: TIME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Tennessee, Knoxville (Other)
Responsible Party: Principal Investigator, Hollie Raynor, Principal Investigator, The University of Tennessee, Knoxville
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UTK_9560 B
Record Dates: First submitted 2014-07-28; First posted 2014-07-30 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2018-04

CONDITIONS: Overweight; Obesity; Weight Loss
Keywords: Meal Time; Weight Loss; Circadian Rhythm
MeSH Terms: conditions — Overweight; Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MORNING (Experimental): Participants will be instructed to consume 50% of their energy intake in their first eating bout, 30% in their second eating bout, and 20% in their third eating bout. For example, a participant prescribed a 1200 kcal/d diet needs to consume 600 kcal in their first eating bout, 360 kcal in their second bout, and 240 kcal in their third bout. Participants will be provided with sample meal plans meeting this prescription.
  Interventions: Behavioral: Eat majority of calories in the morning
- EVENING (Experimental): Participants will be instructed to consume 20% of their energy intake in their first eating bout, 30% in their second eating bout, and 50% in their third eating bout. For example, a participant prescribed a 1200 kcal/d diet needs to consume 240 kcal in their first eating bout, 360 kcal in their second bout, and 600 kcal in their third bout. Participants will be provided with sample meal plans meeting this prescription.
  Interventions: Behavioral: Eat the majority of calories in the evening

INTERVENTIONS:
Behavioral: Eat majority of calories in the morning
  Arms: MORNING
Behavioral: Eat the majority of calories in the evening
  Arms: EVENING

SUMMARY:
While eating the majority of energy earlier in the day appears to have a positive effect on weight and cardiometabolic outcomes, it is not clear how eating earlier in the day influences other behaviors that have a circadian rhythm (sleep), other energy balance behaviors important for weight loss (physical activity), and self-reported feelings of appetite control (hunger and fullness). Thus the purpose of this study is to examine the influence of timing of eating on sleep patterns, physical activity, and self-reported feelings of appetite control. It is hypothesized that those who eat the majority of their calories earlier in the day will have greater weight loss than those who eat the majority later in the day.

DETAILED DESCRIPTION:
Thirty adults will be provided an 8-week standard lifestyle intervention, that includes a 1200-1500 kcal/day, < 30% energy from fat dietary prescription, and a physical activity goal of 200 minutes/week. Participants will be randomized to one of two conditions differing in timing of energy consumed during eating bouts. Both conditions will limit the number of eating bouts/day to three. Participants will be instructed to eat their first eating bout within one hour of awakening and to consume their second and third eating bouts within five or six hours of their previous bout. Participants will be discouraged from eating at least one hour prior to going to sleep. During the intervention, participants will be instructed to self-monitor the time they wake up, the time of the start of each eating bout, and time they go to bed, as well as foods and beverages, and portion sizes, consumed. One condition will consume more energy earlier in the day (MORNING), thus energy intake will be split amongst the three eating bouts with 50% in the first bout, 30% in the second bout, and 20% in the last bout. The second condition will consume more energy later in the day (EVENING), thus energy intake will be split amongst the three eating bouts with 20% in the first bout, 30% in the second bout, and 50% in the last bout.

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) between 27 and 45 kg/m2
* normal self-reported daily (weekday and weekend) wake-up time between 5 am and 8 am
* normal, self-reported weekend wake-up time within two hours of their normal, self-reported weekday wake-up time
* regularly (at least five nights/week) get at least six total hours of self-reported sleep

Exclusion Criteria:

* report a heart condition, chest pain during periods of activity or rest, or loss of consciousness on the Physical Activity Readiness Questionnaire (PAR-Q)
* report being unable to walk for 2 blocks (1/4 mile) without stopping
* are currently participating in a weight loss program and/or taking weight loss medication or lost > 5% of body weight during the past 6 months
* are diagnosed with type 1 or 2 diabetes
* have had bariatric surgery or are planning to have bariatric surgery within the next 4 months
* intend to move outside of the metropolitan area within the time frame of the investigation
* are pregnant, lactating, < 6 months post-partum, or plan to become pregnant during the investigation
* are taking mediation to aid in sleep
* are shift workers/alternative shift workers that work outside of 7 am and 7 pm
* have a metal allergy (which would prevent the ability of participant to wear the SenseWear® armband from BodyMedia® used in the proposed study).

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
weight | 0 and 8 weeks
  Weight will be assessed by an electronic scale, and height will be assessed using a stadiometer, using standard procedures, with participants wearing light clothing, without shoes. BMI (kg/m2) will be calculated from these measures.

SECONDARY OUTCOMES:
physical activity | 0 and 8 weeks
  the SenseWear® armband from BodyMedia will measure physical activity-related energy expenditure for the course of the study. Energy expenditure will be calculated using the corresponding software. This armband reports physical activity in total minutes and joules expended. Furthermore, this armband reports minutes of physical activity divided into 5 categories: sedentary activities (<1.5 METS), light physical activity (1.5-2.9 METS), moderate activity (3.0-5.9 METS), vigorous activity (6.0-8.9 METS), and very vigorous activity (≥9.0 METS). Minutes of active energy expenditure are also reported, which includes total number of minutes engaged in moderate, vigorous, or very vigorous activity. For each participant, mean minutes of sedentary, light, moderate, and vigorous activity (vigorous activity + very vigorous activity) will be calculated over the course of the 7 days.
sleep | 0 and 8 weeks
  participants will be instructed to wear the SenseWear® armband from BodyMedia® on their upper left arm for 7 days. Participants will be instructed to wear the armband for 23 hours a day for each of the 7-day time frames. The SenseWear® has been shown to be a reliable measurement for total sleep time in both individuals with and without obstructive sleep apnea. The SenseWear® armband recognizes the onset of sleep when there is a drop in the heat flux sensor (arm skin temperature).16 The BodyMedia® software then codes the output from the SenseWear® as either wake or sleep (regardless of sleep stage) binary codes,15 based on manufacturer sleep algorithms.16 The armband reports total minutes of lying down and total minutes wake/sleep during the lying down time, allowing sleep efficiency to be calculated. For each participant, minutes of sleep per 24 hrs and mean sleep efficiency will be calculated from the 7 days of measures.
diet | 0 and 8 weeks
  Energy and macronutrient intake overall and per eating bout will be assessed by 3 day (2 weekdays and 1 weekend) food records. Eating bouts will only be counted if at least 25 kcals were consumed. All foods and beverages, eaten within 1/2 h of the start of a meal, will be counted as a single eating bout. To determine dietary variables, each food record will be entered into the Nutrition Data System for Research (NDS-R) software developed by the Nutrition Coordinating Center, University of Minnesota, Minneapolis, Minnesota.
feelings of hunger and fullness | 0 and 8 weeks
  EMA protocol will be conducted over 7 continuous days using both semi-random and event-contingent sampling. Semi-random sampling will assess consumption cues (i.e. feelings of temptation, fullness, desire to eat, energy level and control over eating), along with feelings of hunger, satiation, and deprivation. Event-based sampling will assess these same cues and feelings, as well as reasons for initiating and terminating eating, Time-based and event-based sampling questions will be programmed and displayed using Satellite Forms™ MobileApp Designer software (Thacker Network Technologies Inc., Alberta, Canada).

CONTACTS AND LOCATIONS:
Overall Officials: Hollie Raynor, Ph, RD, Principal Investigator — University of Tennessee
Locations (1):
- Univeristy of Tennessee--HEAL Lab, Knoxville, Tennessee, United States

REFERENCES:
- See also: HEAL research information website — http://nutrition.utk.edu/heal-research/